CLINICAL TRIAL: NCT00861601
Title: TPL111913, a Multi-centre, Open Label, Dose Ranging Phase II Study to Assess Efficacy, Safety and Pharmacokinetics of Eltrombopag in Japanese Thrombocytopenic Subjects With Chronic Liver Disease
Brief Title: Phase 2, Pharmacokinetics Study of Eltrombopag in Japanese Thrombocytopenic Subjects With Chronic Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111913
Record Dates: First submitted 2009-03-05; First posted 2009-03-13 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2011-02

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Tablets; eltrombopag

ARMS (3):
- low dose (Experimental): eltrombopag 12.5 mg/day
  Interventions: Drug: eltrombopag 12.5 milligrams (mg) tablet
- middle dose (Experimental): eltrombopag 25 mg/day
  Interventions: Drug: eltrombopag 25 mg tablet
- high dose (Experimental): eltrombopag 37.5 mg/day
  Interventions: Drug: eltrombopag 12.5 milligrams (mg) tablet; Drug: eltrombopag 25 mg tablet

INTERVENTIONS:
Drug: eltrombopag 12.5 milligrams (mg) tablet — eltrombopag 12.5 mg tablet once a day
  Arms: high dose; low dose
Drug: eltrombopag 25 mg tablet — eltrombopag 25 mg tablet once a day
  Arms: high dose; middle dose

SUMMARY:
This is an open label, multi-centre, dose ranging study to assess efficacy, safety and pharmacokinetics of eltrombopag in thrombocytopenic subjects with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject who agree to comply with protocol requirements and instructions and who provide signed and dated written informed consent.
* Male and female subjects, ≥20 years of age (at the time of informed consent) with chronic liver disease.
* Child-Pugh score <=9.
* A baseline platelet count <50,000/mcL.
* A baseline serum sodium level >130 mEq/L.
* Haemoglobin concentration >8 g/dL, stable for at least 4 weeks.
* A female is eligible to enter and participate in the study if she is of:

Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

* Has had a hysterectomy
* Has had a bilateral oophorectomy (ovariectomy)
* Has had a bilateral tubal ligation
* Is post-menopausal (demonstrate total cessation of menses for longer than one year)

Childbearing potential, has a negative urine and/or serum pregnancy test at screening, and within the 24 hour period prior to the first dose of investigational product and uses one of the following acceptable methods of contraception:

* Complete abstinence from intercourse.
* Any intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Double-barrier contraception (condom with spermicidal jelly, or diaphragm with spermicide).
* Male partner who is sterile (diagnosed by a qualified medical professional) prior to the female subject's study entry and is the sole sexual partner for that female.
* Oral contraceptive (combined).
* Subject has no physical limitation to ingest and retain oral medication.

Exclusion Criteria:

* Subjects with known or suspected hypersensitivity, intolerance or allergy to any of the ingredients in eltrombopag tablets.
* Evidence of portal vein thrombosis on abdominal imaging (ultrasound with Doppler or appropriate magnetic resonance imaging/computed tomography (MRI/CT) imaging techniques) within 3 months before the start of the study.
* History of arterial or venous thrombosis (including Budd-Chiari Syndrome),

AND ≥ two of the following risk factors:

* hereditary thrombophilic disorders (e.g. antithrombinIII (ATIII) deficiency, etc.)
* hormone replacement therapy
* systemic contraception therapy (containing oestrogen)
* smoking
* diabetes
* hypercholesterolemia
* medication for hypertension or cancer
* Human Immunodeficiency Virus (HIV) infection.
* History of drug/alcohol abuse or dependence within 1 year prior to screening.
* Any disease condition associated with current active World Health Organization (WHO) Grade 3 or 4 bleeding.
* Active infection requiring systemic antibiotic therapy.
* Pregnant, nursing mothers, women who may be pregnant, or women who plan to become pregnant during the time of study participation.
* Treatment with platelet transfusion within 2 weeks prior to Day 1.
* Treatment with interferon within 4 weeks prior to Day 1.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* History of platelet agglutination abnormality.
* History of porphyria.
* Subjects who are deemed unsuitable for the study by the investigator (or subinvestigator).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (5):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Ōita

REFERENCES:
- [Background] Kawaguchi T, Komori A, Seike M, Fujiyama S, Watanabe H, Tanaka M, Sakisaka S, Nakamuta M, Sasaki Y, Oketani M, Hattori T, Katsura K, Sata M. Efficacy and safety of eltrombopag in Japanese patients with chronic liver disease and thrombocytopenia: a randomized, open-label, phase II study. J Gastroenterol. 2012 Dec;47(12):1342-51. doi: 10.1007/s00535-012-0600-5. Epub 2012 Jun 8. PMID 22674141

RESULTS

PARTICIPANT FLOW:
Groups:
- Eltrombopag 12.5 mg: Participants received 12.5 milligrams (mg) of eltrombopag once daily for 14 days.
- Eltrombopag 25 mg: Participants received 25 mg of eltrombopag once daily for 14 days. Participants with a platelet count <80 x 10^9/Liter on Day 15 received eltrombopag for an additional week if the participant agreed to it and the investigator considered it appropriate.
- Eltrombopag 37.5 mg: Participants received 37.5 mg of eltrombopag once daily for 14 days. Participants with a platelet count <80 x 10^9/Liter on Day 15 received eltrombopag for an additional week if the participant agreed to it and the investigator considered it appropriate.
Period: Overall Study
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Started | 12 | 14 | 12
Completed | 12 | 14 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg | Total
Number analyzed (Participants) | 12 | 14 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.51) | 57.7 (8.69) | 66.3 (8.84) | 61.8 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 8 | 10 | 8 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese Heritage | 12 | 14 | 12 | 38
Number of participants categorized into the indicated Child-Pugh (CP) Class [Number; unit: participants] — The CP score (ranging from 5 to 15, with 5 being mild and 15 being severe), calculated based on total bilirubin, serum albumin, international normalized ratio, ascites, and hepatic encephalopathy, is used to assess the severity of liver disease. A CP score of 5 or 6 is classified as Class A (mild), a score of 7-9 is classified as Class B (moderate), and a score >=10 is classified as Class C (severe). Participants with a CP score <10 were enrolled in the study
  participants
    Class A | 8 | 8 | 7 | 23
    Class B | 4 | 6 | 5 | 15
    Class C | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Platelet Counts on Day 15
Description: Platelet counts were measured by blood draw. Change from Baseline was calculated as the Day 15 value minus the Baseline value.
Time Frame: Baseline, Day 15
Population: Full Analysis Set (FAS): all enrolled participants, excluding those who received no doses of eltrombopag during the treatment period, those without a baseline platelet assessment, and those without at least one on-therapy (scheduled or unscheduled) platelet assessment.
Measure: Mean (95% Confidence Interval); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter | 24.8 [8.2 to 41.4] | 54.0 [28.2 to 79.8] | 60.0 [29.3 to 90.7]

2. Secondary Outcome: Analysis of Covariance for Three Patterns of Dose Response Using the Change From Baseline in Platelet Counts (Baseline Platelet Counts as Covariate)
Description: Exploratory analysis was conducted to see a dose response/trend when a dose goes high with the changes from baseline in platelet counts (12.5 mg, 25 mg, and 37.5 mg) on Day 15 of each subject. The data were analyzed with baseline of platelet counts as covariate for the following dose response pattern using contrast: (1) linearity, (2) saturation at the medium dose, (3) onset of response at the high dose.
Time Frame: Baseline, Day 15
Population: FAS
Measure: Mean (95% Confidence Interval); unit: 10^9/Liter
Groups:
- Eltrombopag 12.5 mg: Participants received 12.5 mg of eltrombopag once daily for 14 days.
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter | 24.8 [8.2 to 41.4] | 54.0 [28.2 to 79.8] | 60.0 [29.3 to 90.7]
Statistical Analysis 1: Comparison: Eltrombopag 12.5 mg vs Eltrombopag 25 mg vs Eltrombopag 37.5 mg; Test type: Superiority or Other; p = 0.0104, ANCOVA — Linearity. This analysis is based on each participants' change in platelet count; No adjustment for multiplicity was made because this analysis was exploratory
Statistical Analysis 2: Comparison: Eltrombopag 12.5 mg vs Eltrombopag 25 mg vs Eltrombopag 37.5 mg; Test type: Superiority or Other; p = 0.0057, ANCOVA — Saturation at the medium dose. This analysis is based on each participants' change in platelet count; No adjustment for multiplicity was made because this analysis was exploratory
Statistical Analysis 3: Comparison: Eltrombopag 12.5 mg vs Eltrombopag 25 mg vs Eltrombopag 37.5 mg; Test type: Superiority or Other; p = 0.0808, ANCOVA — Onset of response at the higher dose. This analysis is based on each participants' change in platelet count; No adjustment for multiplicity was made because this analysis was exploratory

3. Secondary Outcome: Analysis of Covariance for Three Patterns of Dose Response Using the Change From Baseline in Platelet Counts (Baseline of Platelet Counts and Child-Pugh Class as Covariates)
Description: Exploratory analysis was conducted to see a dose response/trend when a dose goes high with the changes from baseline in platelet counts (12.5 mg, 25 mg, and 37.5 mg) on Day 15 of each subject. The data were analyzed with baseline of platelet counts and Child-Pugh class as covariate for the following dose response pattern using contrast: (1) linearity, (2) saturation at the medium dose, (3) onset of response at the high dose.
Time Frame: Baseline, Day 15
Population: FAS
Measure: Mean (95% Confidence Interval); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter | 24.8 [8.2 to 41.4] | 54.0 [28.2 to 79.8] | 60.0 [29.3 to 90.7]
Statistical Analysis 1: Comparison: Eltrombopag 12.5 mg vs Eltrombopag 25 mg vs Eltrombopag 37.5 mg; Test type: Superiority or Other; p = 0.0116, ANCOVA — Linearity. This analysis is based on each participants' change in platelet count; No adjustment for multiplicity was made because this analysis was exploratory
Statistical Analysis 2: Comparison: Eltrombopag 12.5 mg vs Eltrombopag 25 mg vs Eltrombopag 37.5 mg; Test type: Superiority or Other; p = 0.0066, ANCOVA — Saturation at the medium dose. This analysis is based on each participants' change in platelet count; No adjustment for multiplicity was made because this analysis was exploratory
Statistical Analysis 3: Comparison: Eltrombopag 12.5 mg vs Eltrombopag 25 mg vs Eltrombopag 37.5 mg; Test type: Superiority or Other; p = 0.0846, ANCOVA — Onset of response at the higher dose. This analysis is based on each participants' change in platelet count; No adjustment for multiplicity was made because this analysis was exploratory

4. Secondary Outcome: Percent Change From Baseline in Platelet Counts on Day 15
Description: as for outcome 1
Time Frame: Baseline, Day 15
Population: FAS
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
Percent change | 57.86 [18.77 to 96.94] | 134.57 [81.36 to 187.78] | 158.45 [92.32 to 224.59]

5. Secondary Outcome: Platelet Counts by Treatment Visit
Description: Platelet counts were measured by blood draw. The Final Assessment Point is the last visit during the treatment period, which is Day 15 or Day 22.
Time Frame: Day 1 (Baseline), Day 8, Day 15, and Final Assessment Point (Day 15 or Day 22)
Population: FAS. The number of participants analyzed varies by visit, because the platelet count data on 4 days post-treatment in one participant in the 37.5 mg group are missing and the platelet count data post-specific therapies affecting the evaluation of efficacy are excluded from this efficacy analysis.
Measure: Median (Full Range); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter
  Day 1 | 42.5 [36 to 49] | 38.0 [19 to 48] | 40.0 [23 to 49]
  Day 8 | 50.5 [37 to 73] | 49.5 [27 to 88] | 52.0 [32 to 87]
  Day 15 | 66.0 [37 to 126] | 73.0 [31 to 232] | 81.5 [53 to 242]
  Final Assessment Point | 66.0 [37 to 126] | 95.5 [35 to 232] | 85.5 [57 to 242]

6. Secondary Outcome: Platelet Counts by Post-Treatment Visit
Description: Platelet counts were measured by blood draw.
Time Frame: 4 days post-treatment, 8 days post-treatment, and 15 days post-treatment
Population: as for outcome 5
Measure: Median (Full Range); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 13 | 12
10^9/Liter
  4 days post-treatment, n=12, 13, 11 | 63.5 [41 to 173] | 100.0 [38 to 271] | 109.0 [59 to 372]
  8 days post-treatment, n=12, 13, 12 | 67.5 [46 to 178] | 119.0 [40 to 387] | 120.0 [66 to 376]
  15 days post-treatment, n=11, 13, 11 | 65.0 [36 to 157] | 87.0 [29 to 382] | 97.0 [59 to 295]

7. Secondary Outcome: Platelet Counts at Day 22
Description: as for outcome 5
Time Frame: Day 22
Population: FAS. Participants in the 12.5 mg group have no data on Day 22 because they received the medication for only 14 days. Only 6 participants in the 25 mg group and 2 participants in the 37.5 mg group received the medication for an additional week, because they had a platelet count <80 x 10^9/Liter on Day 15.
Measure: Median (Full Range); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 0 | 6 | 2
10^9/Liter |  | 82.5 [35 to 126] | 72.5 [57 to 88]

8. Secondary Outcome: Change From Baseline in Platelet Counts by Treatment Visit
Description: Platelet counts were measured by blood draw. The Final Assessment Point is the last visit during the treatment period, which is Day 15 or Day 22. Change from Baseline was calculated as the value at each visit minus the Baseline value.
Time Frame: Baseline, Day 8, Day 15, and Final Assessment Point (Day 15 or Day 22)
Population: FAS. The number of participants analyzed varies by visit, because the platelet count data on 4 days post-treatment in one participant in the 37.5 mg group is missing and the platelet count data post-specific therapies affecting the evaluation of efficacy are excluded from this efficacy analysis.
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter
  Day 8 | 6.9 (9.43) | 14.6 (11.80) | 15.4 (8.96)
  Day 15 | 24.8 (26.13) | 54.0 (44.70) | 60.0 (48.36)
  Final Assessment Point | 24.8 (26.13) | 64.0 (42.51) | 61.9 (47.77)

9. Secondary Outcome: Change From Baseline in Platelet Counts by Post-Treatment Visit
Description: Platelet counts were measured by blood draw. Change from Baseline was calculated as the value at each visit minus the Baseline value.
Time Frame: 4 days post-treatment, 8 days post-treatment, and 15 days post-treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 13 | 12
10^9/Liter
  4 days post-treatment, n=12, 13, 11 | 33.0 (36.36) | 73.8 (50.14) | 97.6 (83.38)
  8 days post-treatment, n=12, 13, 12 | 41.5 (40.50) | 100.9 (81.96) | 108.3 (81.26)
  15 days post-treatment, n=11, 13, 11 | 35.7 (36.58) | 82.2 (83.13) | 83.0 (68.31)

10. Secondary Outcome: Percentage of Responders on Day 15
Description: A responder was defined as a participant with a platelet count within the target range (>=80 x 10^9/Liter) on Day 15.
Time Frame: Day 15
Population: FAS
Measure: Mean (95% Confidence Interval); unit: percentage of responders
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
percentage of responders | 25.0 [5.5 to 57.2] | 42.9 [17.7 to 71.1] | 58.3 [27.7 to 84.8]

11. Secondary Outcome: Percentage of Responders on Day 22
Description: A responder was defined as a participant with a platelet count within the target range (>=80 x 10^9/Liter) on Day 22 after receiving eltrombopag for an additional week from Day 15, on which his or her platelet count was <80 x 10^9/Liter.
Time Frame: Day 22
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: percentage of responders
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 0 | 6 | 2
percentage of responders |  | 50.0 [11.8 to 88.2] | 50.0 [1.3 to 98.7]

12. Secondary Outcome: Change From Baseline in Platelet Counts on Day 15 by Child-Pugh Class
Description: Change from Baseline was calculated as the Day 15 value minus the Baseline value. The Child-Pugh (CP) score (ranging from 5 to 15, with 5 being mild and 15 being severe), calculated based on total bilirubin, serum albumin, international normalized ratio, ascites, and hepatic encephalopathy, is used to assess the severity of liver disease. A CP score of 5 or 6 is classified as Class A (mild), a score of 7-9 is classified as Class B (moderate), and a score >=10 is classified as Class C (severe). Participants with a CP score <10 were enrolled in the study.
Time Frame: Baseline, Day 15
Population: FAS. The number of participants categorized as Class A or Class B is given in the category titles.
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter
  Child-Pugh Class A, n=8, 8, 7 | 24.4 (32.51) | 44.5 (27.02) | 66.6 (60.59)
  Child-Pugh Class B, n=4, 6, 5 | 25.8 (5.97) | 66.7 (61.93) | 50.8 (27.23)

13. Secondary Outcome: Change From Baseline in Platelet Counts on Day 15 by Sex
Description: Change from Baseline was calculated as the Day 15 value minus the Baseline value. The numbers of females and males in each treatment group are illustrated by the "n's" in the category titles.
Time Frame: Baseline, Day 15
Population: FAS
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter
  Female, n=4, 4, 4 | 47.3 (31.16) | 83.5 (69.67) | 98.8 (65.18)
  Male, n=8, 10, 8 | 13.6 (15.03) | 42.2 (26.96) | 40.6 (23.81)

14. Secondary Outcome: Change From Baseline in Platelet Counts on Day 15 by Age
Description: Change from Baseline was calculated as the Day 15 value minus the Baseline value. The numbers of participants in each age category are illustrated by the "n's" in the category titles.
Time Frame: Baseline, Day 15
Population: FAS
Measure: Mean (Standard Deviation); unit: 10^9/Liter
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Number analyzed (Participants) | 12 | 14 | 12
10^9/Liter
  <65 years of age, n=7, 11, 5 | 19.7 (23.34) | 40.2 (24.50) | 49.8 (30.36)
  >=65 years of age, n=5, 3, 7 | 32.0 (30.82) | 104.7 (71.32) | 67.3 (59.36)

15. Secondary Outcome: Log-transformed Cmax on Days 14 and 15 in Participants Receiving Eltrombopag 12.5 mg
Description: Serial PK samples were collected over a 24-hour (h) period on Days 14 and 15 in participants receiving eltrombopag 12.5 mg. A total of 8 blood samples (3 milliliters per sample) were collected at pre-dose, and at 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, and 24 h post-dose. Cmax=maximum drug concentration.
Time Frame: Day 14, Day 15
Population: PK Parameter Population: all participants from whom a PK sample was obtained and analyzed and whose PK parameter data was evaluated. One of the 12 participants took a prohibited medication that might have decreased the absorption of eltrombopag during the treatment period and was hence excluded from the PK Parameter Population.
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms/milliliter (ng/ml)
Arm/Group | Eltrombopag 12.5 mg
Number analyzed (Participants) | 11
nanograms/milliliter (ng/ml) | 3412.999 [2549.0060 to 4569.8448]

16. Secondary Outcome: Log-transformed Tmax on Days 14 and 15 in Participants Receiving Eltrombopag 12.5 mg
Description: Serial PK samples were collected over a 24-hour (h) period on Days 14 and 15 in participants receiving eltrombopag 12.5 mg. A total of 8 blood samples (3 milliliters per sample) were collected at pre-dose, and at 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, and 24 h post-dose. Tmax=maximum drug concentration time.
Time Frame: Day 14, Day 15
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Eltrombopag 12.5 mg
Number analyzed (Participants) | 11
hours | 3.444 [2.4593 to 4.8226]

17. Secondary Outcome: Log-transformed AUC(0-t) and AUC(0-24) on Days 14 and 15 in Participants Receiving Eltrombopag 12.5 mg
Description: Serial PK samples were collected over a 24-hour (h) period on Days 14 and 15 in participants receiving eltrombopag 12.5 mg. A total of 8 blood samples (3 milliliters per sample) were collected at pre-dose, and at 1 h, 2 h, 4 h, 6 h, 8 h, 10 h, and 24 h post-dose. AUC(0-t)=area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration, and AUC(0-24)=area under the concentration-time curve from 0 (pre-dose) to 24 hours.
Time Frame: Day 14, Day 15
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hours * ng/ml
Arm/Group | Eltrombopag 12.5 mg
Number analyzed (Participants) | 11
hours * ng/ml
  AUC(0-t) | 65244.180 [46617.4188 to 91313.5730]
  AUC(0-24) | 65235.699 [46748.123 to 91034.594]

ADVERSE EVENTS:
Time Frame: The time period of detecting adverse events (AEs) and serious adverse events (SAEs) was from the start of eltrombopag (Day 1) treatment to 15 days post-treatment.
Arm/Group | Eltrombopag 12.5 mg | Eltrombopag 25 mg | Eltrombopag 37.5 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 1/12
Other Adverse Events (participants affected / at risk) | 6/12 | 7/14 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag 12.5 mg (N=12) | Eltrombopag 25 mg (N=14) | Eltrombopag 37.5 mg (N=12)
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag 12.5 mg (N=12) | Eltrombopag 25 mg (N=14) | Eltrombopag 37.5 mg (N=12)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 2
Malaise (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 3 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Renal disorder (Renal and urinary disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.